CLINICAL TRIAL: NCT03798249
Title: Effect of Acute and Sub-acute Administration of Gluten on Extra-intestinal and Gastrointestinal Symptoms in Patients With Non-coeliac Gluten Sensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: S60127
Record Dates: First submitted 2018-10-11; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: NCGS; Gluten
MeSH Terms: interventions — Glutens

STUDY DESIGN:
Intervention Model Description: single-blinded, randomised - controlled, crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten (Active Comparator): Patients will receive acutely 16 g of gluten and 2 muffins glutenfree with 8 g of gluten, twice a day, during 5 days
  Interventions: Other: Gluten
- Placebo (Placebo Comparator): Patients will receive acutely 16 g of whey protein and 2 glutenfree muffins, twice a day, during 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Gluten — Tereos
  Arms: Gluten
Other: Placebo — Nestlé Health Science
  Arms: Placebo

SUMMARY:
The investigators will investigate the effects of acute and sub-acute administration of gluten on mood, intestinal permeability, gastrointestinal symptoms, gut microbiota and cortisol levels in NCGS patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-coeliac gluten sensitivity patients

  * Previous symptoms of IBS fulfilling Rome III criteria that self reportedly improved with a gluten-free diet
  * Symptoms currently well controlled on a gluten-free diet
  * Adherence to the gluten-free diet for at least 6 weeks prior to recruitment
  * Coeliac disease excluded (either by absence of the HLA-DQ2 and HLA-DQ8 haplotype or by a normal duodenal biopsy (Marsh 0) performed at endoscopy while on a gluten-containing diet in individuals expressing the HLA-DQ2 or HLA-DQ8 haplotype)
  * IgA anti-tissue-transglutaminase or IgG anti-deaminated gliadin peptide positive
* Body Mass Index (BMI) of 20 - 25 kg/m2
* Stable body weight for at least 3 months prior to the start of the study

Exclusion Criteria:

* Medical

  * Coeliac disease
  * Abdominal or thoracic surgery. Exception: appendectomy
  * Gastrointestinal, endocrine or neurological diseases
  * Cardiovascular, respiratory, renal or urinary diseases
  * Hypertension
  * Food or drug allergies
* Psychiatric disorders

  * Eating disorders
  * Depressive disorders
  * Anxiety disorders
  * Psychotic disorders
* Restraint or emotional eating
* Medication on a regular basis, exception: oral contraception
* History of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Alcohol abuse (more than 21 units of alcohol for men, more than 14 units for woman per week)
* Pregnant or breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The effect of gluten acutely and sub-acutely on extraintestinal symptoms in NCGS patients measured on the Positive and Negative Affect Schedule | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 20), after test visit 3 (at day 35), after test visit 4 (at day 40)
  Change from baseline. Scores can be 'very slightly or not at all', 'a little', 'moderately', 'quite a bit', 'extremely'
The effect of gluten acutely and sub-acutely on extraintestinal symptoms in NCGS patients measured on the Profile of Mood State | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 20), after test visit 3 (at day 35), after test visit 4 (at day 40)
  Scores are measured on the Visual Analogue Scale. Change from baseline. The scale is ranged 0 - 10, in which 0 no occurrence of the symptom and 10 a lot occurrence of the symptom. Measured at day 0, day 15, day 21, day 36 and day 41.

SECONDARY OUTCOMES:
The effect of gluten acutely and sub-acutely on gastrointestinal symptoms in NCGS patients measured on the visual analogue scale for gastrointestinal symptoms | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 20), after test visit 3 (at day 35), after test visit 4 (at day 40)
  With '0' no complaints and '10' a lot of complaints (change from baseline). Measured on the Visual Analogue Scale. Measured at day 0, day 15, day 21, day 36 and day 41.
Effect of acute and sub-acute gluten administration on intestinal permeability (lactulose mannitol ratio) | At the beginning of test visit 0 (day 0), visit 1 (at day 15), test visit 2 (at day 21), after test visit 3 (at day 36), after test visit 4 (at day 41)
  Change in intestinal permeability after gluten administration. In the urine we can measure the ratio lactulose/mannitol. This can be measured using High Performance Liquid Chromatography at day 0, day 15, day 21, day 36 and day 41.
Effect of acute and sub-acute gluten administration on high sensitive reactive protein levels in bloodsample | During test visit 0 (day 0), test visit 2 (at day 21), after test visit 4 (at day 41)
  Change in high sensitive reactive protein levels measured at day 0, day 21 and day 41
Effect of acute and sub-acute gluten administration on Lipopolysaccharide-Binding Protein levels in bloodsample | During test visit 0 (day 0), test visit 2 (at day 21), after test visit 4 (at day 41)
  Change in lipopolysaccharide-binding protein levels measured at day 0, day 21 and day 41
Effect of acute and sub-acute gluten administration on lipopolysaccharide levels in bloodsample | During test visit 0 (day 0), test visit 2 (at day 21), after test visit 4 (at day 41)
  Change in lipopolysaccharide levels measured at day 0, day 21 and day 41
Effect of acute and sub-acute gluten administration on gut microbiota composition | After test visit 0 (day 0), day 13 and day 14, after test visit 1 (day 15), day 16, 17, 18, 19 and 20, two days before test visit 3 (day 34 and 35), day 36, 37, 38, 39, 40
  Change in gut microbiota composition (compared to day 0) with focus on: Bifidobacterium, Lactobacillus, Enterobacteriaceae, E. coli (stool samples)
Effect of acute and sub-acute gluten administration on cortisol awakening response | Day before test visit 1 (day 14), test visit 1 (day 15), test visit 2 (day 21), day before test visit 3 (day 35), test visit 3 (day 36) and test visit 4 (day 41)
  Change in cortisol levels between gluten and placebo administration (saliva samples). Measured using an ELISA assay.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - TARGID, Leuven, Vlaams-Brabant
  - Jan Tack, Leuven

REFERENCES:
- [Derived] Iven J, Geeraerts A, Vanuytsel T, Tack J, Van Oudenhove L, Biesiekierski JR. Impact of Acute and Sub-Acute Gluten Exposure on Gastrointestinal Symptoms and Psychological Responses in Non-Coeliac Gluten Sensitivity: A Randomised Crossover Study. United European Gastroenterol J. 2025 Sep;13(7):1295-1306. doi: 10.1002/ueg2.70014. Epub 2025 Mar 26. PMID 40138597